CLINICAL TRIAL: NCT03778281
Title: Open-label Randomized Controlled Prospective Study of Baclofen in the Treatment of Chemotherapy-related Hiccups
Brief Title: Treatment of Chemotherapy-related Hiccups With Baclofen
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HL002
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Hiccup
Keywords: Baclofen; Chemotheropy
MeSH Terms: conditions — Hiccup | interventions — Baclofen; Inactivation, Metabolic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient privacy needs to be protected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baclofen group (Experimental): Treatment of Chemotherapy-related Hiccups With Baclofen
  Interventions: Drug: Baclofen
- Methoxyclopramide group (Other): Treatment of Chemotherapy-related Hiccups With Methoxyclopramide
  Interventions: Drug: Methoxyclopramide
- Baclofen group 2 (Experimental): After 3 days, if the metoclopramide treatment is ineffective, it will cross into the baclofen group 2.
  Interventions: Drug: Baclofen
- Methoxyclopramide group 2 (Other): After 3 days, if the baclofen treatment is ineffective, it will cross into the metoclopramide group 2.
  Interventions: Drug: Methoxyclopramide

INTERVENTIONS:
Drug: Baclofen — Oral baclofen 10mg, 3 times a day for three days, then evaluate the efficacy and side effects
  Other Names: Baclofenum、Gabalon、Lioresal
  Arms: Baclofen group; Baclofen group 2
Drug: Methoxyclopramide — Intramuscular injection of metoclopramide 10mg, 3 times a day for three days, then evaluate the efficacy and side effects
  Other Names: Detoxification
  Arms: Methoxyclopramide group; Methoxyclopramide group 2

SUMMARY:
Hiccup is one of the common side effects of chemotherapy. Intractable hiccups seriously affect patients' rest and eating, reduce the quality of life, and increasingly attract the attention of oncologists. At present, drugs or methods for treating chemotherapy-related hiccups are generally ineffective, with short remission time, serious adverse reactions, and unsatisfactory clinical effects. Baclofen produces skeletal muscle relaxation and was originally used in patients with spinal cord injury, and has since been used to treat intractable hiccups caused by diaphragmatic spasm. This study was an open-label, randomized, prospective study comparing the efficacy and adverse effects of baclofen versus metoclopramide in the treatment of chemotherapy-related hiccups. Patients with hiccup after chemotherapy were randomly divided into two groups. One group was treated with baclofen and the other group was treated with metoclopramide. The efficacy and adverse reactions of the two groups were compared.Ineffective in the two groups will cross to another group and then observe the efficacy.

DETAILED DESCRIPTION:
Hiccup is due to paroxysmal paralysis of the diaphragm, sudden inhalation of gas accompanied by rapid glottis closure and a short high-pitched sound, commonly known as "snoring", is one of the common adverse reactions of chemotherapy. Intractable hiccups seriously affect the rest and eating of patients, reduce the quality of life, and increasingly attract the attention of oncologists. At present, the drugs or methods used in the treatment of chemotherapy-related hiccups mainly include chlorpromazine, Ritalin, diazepam, phenacetin, metoclopramide and traditional Chinese medicine, but these drugs or treatments usually have poor efficacy and short remission time. The adverse reactions were serious and the clinical use was not satisfactory. Baclofen is a gamma-aminobutyric acid (GABA) derivative that activates the GABA-β receptor, inhibits the release of excitatory neurotransmitters, and reduces monosynaptic or multisynaptic transmission in the spinal cord. Skeletal muscle relaxation, originally used in patients with spinal cord injury, is gradually used to treat intractable hiccups caused by diaphragmatic spasm.

This study was an open-label, randomized, prospective study comparing the efficacy and adverse effects of baclofen versus metoclopramide in the treatment of chemotherapy-related hiccups. Patients with hiccup after chemotherapy were randomly divided into two groups. One group was treated with baclofen and the other group was treated with metoclopramide. The efficacy and adverse reactions of the two groups were compared.Ineffective in the two groups will cross to another group and then observe the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of malignant tumors;PS score 0 ~ 3 points;
* Hiccups occurred within 48 h after chemotherapy, lasting longer than 2 h.

Exclusion Criteria:

* No serious heart, brain, lung, kidney and other diseases, no gastrointestinal bleeding, no serious obstacles to blood clotting;
* Blood routine and normal electrolyte of liver and kidney function before chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-12-12 (Estimated); Primary Completion 2019-12-11 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Effective rate | 3 days
  Effective rate includes complete response rate and partial response rate

SECONDARY OUTCOMES:
Adverse reactions | 3 days
  Adverse reactions include drowsiness, dizziness, sedation, tremors, etc.

CONTACTS AND LOCATIONS:
Overall Officials: long Huang, Phd, Study Director — Second Affiliated Hospital of Nanchang University

IPD SHARING:
Plan to Share IPD: No